CLINICAL TRIAL: NCT07394036
Title: The Effect of Ipratropium Bromide on Exercise-Induced Laryngeal Obstruction (EILO) in Pediatric Patients
Brief Title: Effect of Ipratropium Bromide on EILO
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cook Children's Health Care System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025-042
Record Dates: First submitted 2026-01-12; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Exercise-Induced Laryngeal Obstruction; Dyspnea During Activity
Keywords: Exercise-Induced Laryngeal Obstruction; Shortness of Breath during Exercise; Ipratropium Bromide
MeSH Terms: interventions — Ipratropium; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ipratropium Bromide, then Placebo (Experimental): Participants will receive Ipratropium Bromide in their first trial and Placebo in the second trial.
  Interventions: Drug: Ipratropium Bromide; Drug: Normal Saline (Placebo)
- Placebo, then Ipratropium Bromide (Experimental): Participants will receive Placebo in their first trial and Ipratropium Bromide in the second trial.
  Interventions: Drug: Ipratropium Bromide; Drug: Normal Saline (Placebo)

INTERVENTIONS:
Drug: Ipratropium Bromide — Nebulized Ipratropium Bromide (500µg/2.5mL); one-time dose approximately 75 minutes before exercise, inhaled for 5-8 minutes
Drug: Normal Saline (Placebo) — 3 mL of nebulized 0.9% normal saline; one-time dose approximately 75 minutes before exercise, inhaled for 5-8 minutes

SUMMARY:
The investigators propose a study that compares breathlessness and airway obstruction during intense exercise in 34 children and adolescents with Exercise-Induced Laryngeal Obstruction after breathing in ipratropium bromide or placebo. It is hypothesized that breathlessness and airway obstruction will be lower following breathing in ipratropium bromide compared with placebo.

DETAILED DESCRIPTION:
Many children and adolescents struggle with breathing problems during exercise. These symptoms can lead them to underperform, quit sports, and in some cases, stop being active altogether. One under-recognized cause is Exercise-Induced Laryngeal Obstruction (EILO), a narrowing of the airway at the level of the voice box. Approximately 5-8% of adolescents and 20-40% of adolescent athletes have EILO, an estimated 4-6 million nationwide. The most common treatment for EILO is Speech Therapy, with or without Physical Therapy. Where available, this requires significant time and financial commitment from patients and their families to attend therapy sessions and complete at-home exercises.

Case reports as early as 1985 have suggested aerosolized ipratropium bromide as an effective EILO treatment. One larger study could not confirm this observation. However, this study used an outcome measure with low reliability and validity, did not use a placebo control, and administered a low dose of ipratropium bromide too close to exercise.

The investigators propose a study that compares breathlessness and airway obstruction during intense exercise in 34 children and adolescents with EILO following inhalation of a higher dose of nebulized ipratropium bromide with placebo. It is hypothesized that breathlessness and airway obstruction will be lower following inhalation of ipratropium bromide compared with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be diagnosed with EILO confirmed by Continuous Laryngoscopy During Exercise
* Patients must be able to complete exercise testing
* Patients must report dyspnea
* Patients must have given assent with parental consent, understand all study procedures, and comply with them for the entire length of the study.

Exclusion Criteria:

* Patients that do not have EILO.
* Patients who did not undergo diagnostic CPET with CLE.
* Patients with hypersensitivity to atropine or its derivatives due to structural similarity with ipratropium bromide.
* Patients with a history of atrial flutter and/or fibrillation
* Patients taking anticholinergic medications that cannot be paused for 24 hours.
* Unable to perform exercise tests
* Current drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Inability or unwillingness of patient or parent/legally authorized representative to give written informed consent.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2026-03-16 (Estimated); Primary Completion 2029-03-30 (Estimated); Study Completion 2029-03-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale for Dyspnea (VAS-Dyspnea) | Day1 and Day 2
  Shortness of breath assessed by a 0-100 Visual Analogue Scale for Dyspnea, where higher scores reflect greater breathlessness

SECONDARY OUTCOMES:
CLE grade scoring | Day 1 and Day 2
  Patient videos will be assessed for laryngeal obstruction by two expert reviewers. Blinded reviewers will grade the severity of glottic and supraglottic obstruction on a scale from 0 (no obstruction) to 3 (severe obstruction).

CONTACTS AND LOCATIONS:
Locations (1):
- Cook Children's Pulmonology (Exercise Respiratory Center), Prosper, Texas, United States

IPD SHARING:
Plan to Share IPD: No
The investigators anticipate the institution's IRB/legal team will not approve sharing IPD.